CLINICAL TRIAL: NCT01807559
Title: SoundBite Hearing System 24 Month Multi Site Patient Use Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sonitus Medical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN009
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Single Sided Deafness; Conductive Hearing Loss
Keywords: Single Sided Deafness; Conductive Hearing Loss; Unilateral Hearing Loss; SSD
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Unilateral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SoundBite Hearing System — The Sonitus Medical SoundBite Hearing System prosthetic device is a bone conduction device that has been FDA cleared for the treatment of single-sided deafness (SSD) and conductive hearing loss (CHL). The Sonitus Medical SoundBite Hearing System consists of an In-the-Mouth (ITM) component, an external microphone component worn behind the ear (BTE), a calibration interface cable and PC-controlled software for subject calibration. A charger is also provided to charge the ITM and the BTE. The objective of this study is multi-site observational study is to asses the long-term patient use of the Sonitus Medical SoundBite Hearing System.

SUMMARY:
The objective of this multi-site observational study is to further assess the long-term patient use of the Sonitus SoundBite Hearing System. Information can be gained by assessing benefit for the subjects that were enrolled in the SoundBite Hearing System Long Term Multi Site Study (Protocol CLN006) for an additional 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who previously were enrolled in SoundBite Hearing System Long Term Multi Site Patient Use Study (Protocol CLN006) and completed the 12 month study visit.
* Additionally, subjects must meet one of the two criteria for hearing loss:

  1. Moderately severe, severe, or profound sensorineural hearing loss in one ear and normal hearing in the other ear (i.e. single sided deafness or "SSD"). Normal hearing is defined as a pure tone average (PTA) air-conduction (AC) hearing threshold (measured at 0.5, 1, 2, and 3 kHz) of better than or equal to 25 dB HL.

     OR
  2. Conductive hearing loss where the pure tone average bone-conduction hearing threshold (measured at 0.5, 1, 2, and 3 kHz) is better than or equal to 25 dB HL.

Exclusion Criteria:

* Subjects that do not meet one of the two the audiometric criteria as measured on the audiogram for the 12 month study appointment for Protocol CLN006:

  1. A moderately severe, severe, or profound sensorineural hearing loss in one ear and normal hearing in the other ear (i.e. single sided deafness or -SSD‖). Normal hearing is defined as a pure tone average (PTA) air-conduction (AC) hearing threshold (measured at 0.5, 1, 2, and 3 kHz) of better than or equal to 25 dB HL.
  2. Patients with conductive hearing loss where the pure tone average bone-conduction hearing threshold (measured at 0.5, 1, 2, and 3 kHz) is better than or equal to 25 dB HL

     * The SoundBite Hearing System and all portions of it are contraindicated for use in an MRI Environment and should be removed prior to MRI exposure
     * The SoundBite Hearing System is not to be used in patients with known hypersensitivity to any of the components including allergies to polymers.
     * The SoundBite Hearing system is contraindicated for vulnerable populations that are unable to use their hands such as paraplegics or others that are unable to comply with the warnings in the product's labeling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All trial subjects are individuals who are already currently using SoundBite Hearing System for treatment of their SSD or CHL and were enrolled in the SoundBite Hearing System Long Term Multi Site Patient Use Study (Protocol CLN0006). Participants are willing to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Abbreviated Profile of Hearing Aid Benefit (APHAB) Questionnaire | 24 Months
  Change in Abbreviated Profile of Hearing Aid Benefit (APHAB, Form A- New Formate, Hearing Aid Research Lab, University of Memphis, 1994) score at 24 months compared to baseline.

SECONDARY OUTCOMES:
Aided Threshold Testing | 24 Months
  Aided Threshold testing of the impaired ear at 24 months as compared with baseline using the SoundBite Hearing System

OTHER OUTCOMES:
Single Sided Deafness Questionnaire | 24 Months
  This questionnaire assesses quality of life outcomes.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Arizona Ear Center, Phoenix, Arizona
  - California Hearing and Balance, La Jolla, California
  - Shohet Ear Associates, Newport Beach, California
  - The George Washington University-Department of Otolaryngology, Washington D.C., District of Columbia
  - Physicians Choice Hearing and Balance, Tampa, Florida
  - Ear Medical Group, San Antonio, Texas
  - University Health Science Center (University of Utah Hospital), Salt Lake City, Utah

REFERENCES:
- See also: Related Info — http://soundbitehearing.com